CLINICAL TRIAL: NCT02409355
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) Compared With Gemcitabine+Cisplatin or Carboplatin for PD-L1-Selected, Chemotherapy Naive Patients With Stage IV Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab Compared With Gemcitabine Plus (+) Cisplatin or Carboplatin for PD-L1-Selected Participants With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC) (IMpower111)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was closed due to low patient enrollment and the Sponsor's decision to include patients with squamous NSCLC into the GO29431 study, NCT02409342.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29432; 2014-003106-33 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Carboplatin; Cisplatin; Gemcitabine

ARMS (2):
- Atezolizumab (Experimental): Participants will receive intravenous (IV) infusion of atezolizumab once on Day 1 of each 21-day cycle until loss of clinical benefit.
  Interventions: Drug: Atezolizumab
- Gemcitabine + Cisplatin/Carboplatin (Active Comparator): Participants will receive IV infusion of gemcitabine + cisplatin or gemcitabine + carboplatin once on Day 1 of each 21-day cycle for four or six cycles as per local standard of care.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 milligrams (mg) by IV infusion on Day 1 of each 21-day cycle until loss of clinical benefit.
  Other Names: MPDL3280A; Tecentriq
  Arms: Atezolizumab
Drug: Carboplatin — Carboplatin will be administered at area under the concentration-time curve (AUC) 5 IV infusion once on Day 1 of each 21-day cycle for 4 or 6 cycles.
  Arms: Gemcitabine + Cisplatin/Carboplatin
Drug: Cisplatin — Cisplatin will be administered at 75 milligrams per square meter (mg/m^2) IV infusion once on Day 1 of each 21-day cycle for 4 or 6 cycles.
  Arms: Gemcitabine + Cisplatin/Carboplatin
Drug: Gemcitabine — Gemcitabine will be administered at 1000 mg/m^2 (when coadministered with carboplatin) or 1250 mg/m^2 (when coadministered with cisplatin) IV infusion on Days 1 and 8 of each 21-day cycle for 4 or 6 cycles.
  Arms: Gemcitabine + Cisplatin/Carboplatin

SUMMARY:
This randomized, open-label study was designed to evaluate and compare the safety and efficacy of atezolizumab with gemcitabine + cisplatin or carboplatin in PD-L1 selected participants with chemotherapy-naive, Stage IV squamous NSCLC. The study was closed due to low patient enrollment and the Sponsor's decision to include patients with squamous NSCLC into the GO29431 study, NCT02409342. Therefore the planned objectives of this study are no longer applicable and formal analyses of efficacy or safety have not been performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IV squamous NSCLC
* Tumor programmed death-ligand 1 (PD-L1) expression, as determined by immunohistochemistry (IHC) assay of archival tumor tissue or tissue obtained at screening
* No prior treatment for Stage IV squamous NSCLC
* Measurable disease as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases
* Untreated or inadequately treated spinal cord compression
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia
* Any other malignancies within 5 years except those with negligible risk of metastasis or death
* Pregnant or lactating women
* Known hypersensitivity to any component of atezolizumab formulation or other study medication
* History of autoimmune disease except controlled, treated hypothyroidism or type I diabetes
* Prior allogeneic bone marrow or solid organ transplantation
* Positive human immunodeficiency virus (HIV) test
* Active hepatitis B or C
* Active tuberculosis
* Significant cardiovascular disease
* Severe infection or major surgery within 4 weeks prior to randomization
* Use of any approved anti-cancer therapy within 3 weeks prior to treatment
* Use of an investigational agent or participation in another clinical trial within 4 weeks prior to randomization
* Exposure to oral or IV antibiotics within 2 weeks or live attenuated vaccines within 4 weeks prior to randomization
* Prior treatment with cluster of differentiation (CD) 137 agonists or immune checkpoint blockade therapies, anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies
* Treatment with immunostimulatory agents within 4 weeks or immunosuppressive agents within 2 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (28):
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - Marin Cancer Care Inc, Greenbrae, California
  - University of California San Diego, La Jolla, California
  - Chao Family Comprehensive Cancer Center; UC Irvine Medical Center, Orange, California
  - Eastern Connecticut Hematology and Oncology Associates; (ECHO), Norwich, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Straub Clinic & Hospital; Oncology, Honolulu, Hawaii
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Consultants in Blood Disorders & Cancer, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - Montana Cancer Specialists, Missoula, Montana
  - Atlantic Health Cancer Center, Summit, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - First Health of the Carolinas, Pinehurst, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Wellmont Cancer Institute, Bristol, Tennessee
  - University Oncology Associates, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Germantown, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Multiscan s.r.o., Pardubice, Czechia
- France (3):
  - Hôpital du Cluzeau, Limoges
  - Hopital Tenon; Oncologie Radiotherapie, Paris
  - Centre Paul Strauss, Strasbourg
- Germany (2):
  - KRH Klinikum Siloah-Oststadt-Heidehaus, Hanover
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
- Greece (4):
  - Sotiria Chest Hospital of Athens, Athens
  - Attikon University General Hospital, Athens
  - Bioclinic Thessaloniki, Thessaloniki
  - Georgios Papanikolaou General Hosp. of Thessaloniki, Thessaloniki
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Matrai Gyogyintezet, Mátraháza
  - Szabolcs-Szatmar-Bereg Megyei; Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Pecs, I st Dept of Internal Medicine, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rend.Int., Szolnok
- Italy (12):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona, Lombardy
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - A.O.U.I. VERONA-OSPEDALE BORGO TRENTO; ONCOLODIA MEDICA-d.O., Verona, Veneto
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- Romania (7):
  - County Hospital Alba; Oncology, Alba Iulia
  - Dr Constantin Opris Emergency County Hospital Baia Mare, Baia Mare
  - Teo Health SA - Saint Constantin Hospital, Brasov
  - Oncology Center Sf. Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi; Clinica de Hematologie, Iași
  - Sibiu Emergency Clinical County Hospital, Sibiu
  - Oncomed SRL, Timișoara
- Russia (5):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - Filial #1 Regional Oncology Dispensary of Nizhniy Novgorod, Nizhny Novgorod
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Mordovia State University, Saransk
- Serbia (3):
  - Clinical Hospital Center Bezanijska kosa; Clinic for Oncology, Belgrade
  - Institute of Lung Diseases Vojvodina, Kamenitz
  - Clin Hospital Center - Kragujevac; Pulmonary Diseases, Kragujevac
- South Korea (3):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Fundacion Investigacion Hospital La Fe de Valencia, Valencia
  - Hosp Clinico Univ Lozano Blesa, Zaragoza
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Diana Princess of Wales Hosp., Grimsby
  - Sarah Cannon Research Institute, London
  - Christie Hospital NHS Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atezolizumab | Gemcitabine + Cisplatin/Carboplatin
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 1
Not completed — Study terminated by Sponsor | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Gemcitabine + Cisplatin/Carboplatin | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time Frame: Baseline up to death or disease progression, whichever occurs first (up to approximately 2.5 years)
Population: The study was closed due to low patient enrollment and the Sponsor's decision to include patients with squamous NSCLC into the GO29431 study. The planned outcome measures of this study are no longer applicable. The outcome measures were removed in the last protocol version.
Arm/Group | Atezolizumab | Gemcitabine + Cisplatin/Carboplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 19 months
Description: Safety Populiation
Arm/Group | Atezolizumab | Gemcitabine + Cisplatin/Carboplatin
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=4) | Gemcitabine + Cisplatin/Carboplatin (N=4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=4) | Gemcitabine + Cisplatin/Carboplatin (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (2)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (2)
PYREXIA (General disorders) | 2 (2) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 0 (0)
DYSMETRIA (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOSIS IN DEVICE (Product Issues) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
GLOMERULONEPHRITIS MEMBRANOUS (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY FIBROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL TUBULAR ATROPHY (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was closed due to low enrollment and the Sponsor's decision to include patients with squamous NSCLC into the GO29431 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT02409355/Prot_SAP_000.pdf